CLINICAL TRIAL: NCT06614738
Title: Microbial and Environmental Factors Associated with Polyps Development in Familial Adenomatous Polyposis
Brief Title: Microbial and Environmental Factors Associated with Polyps Development in Familial Adenomatous Polyposis (MicrobEnvironment in FAP)
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL24_0139; 2024-A01814-43 (Other: Agence nationale de sécurité du médicament et des produits de santé)
Record Dates: First submitted 2024-09-24; First posted 2024-09-26 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Familial Adenomatous Polyposis
Keywords: Familial adenomatous polyposis; microbiota; colorectal cancer; nutrition
MeSH Terms: conditions — Adenomatous Polyposis Coli; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — * Blood sampling (plasmotheque and serotheque): 2 tubes (EDTA (5mL) and dry (5mL)) during hospitalization
  * Fecal sampling (fecal library): A stool sample (approx. 2g) will be taken 48 hours before the endoscopy
  * Duodenal aspiration fluid (6-10 mL in total): before and after mucosal lavage with sterile isotonic saline on the day of endoscopy.
  * Food and Lifestyle Questionnaire (FFQ) during inclusion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with genetically proven familial adenomatous polyposis undergoing surgery: Patients with familial adenomatous polyposis hospitalized for regular endoscopic follow-up by upper and lower digestive endoscopy at Hôpital Edouard Herriot, Lyon, France or Hôpital de la Croix-Rousse, Lyon, France
  Interventions: Other: Sampling of feces and duodenal fluids

INTERVENTIONS:
Other: Sampling of feces and duodenal fluids — * Blood sampling (plasmotheque and serotheque): 2 tubes (EDTA (5mL) and dry (5mL)) during hospitalization
  * Fecal sampling (fecal library): A stool sample (approx. 2g) will be taken 48 hours before the endoscopy at home for outpatient or during hospitalization
  * Duodenal aspiration fluid (6-10 mL in total): before and after mucosal lavage with sterile isotonic saline on the day of endoscopy.
  * Food and Lifestyle Questionnaire (FFQ) during inclusion

SUMMARY:
Familial adenomatous polyposis (FAP) is an autosomal dominant inherited disorder linked to a mutation in the APC gene, associated with the development of multiple colonic and duodenal adenomas, which in 100% of cases progress to colorectal cancer (CRC) if left untreated. Management of affected patients is usually based on prophylactic total colectomy with or without rectal preservation, followed by regular endoscopic surveillance of the duodenum and rectum or ileal reservoir. However, there is considerable inter- and intra-familial variability in the rate of adenoma appearance and development for identical mutations. This strongly suggests the additional role of environmental factors. Recently, the gut microbiota has been identified as a co-factor of carcinogenesis in patients with FAP, but no prospective evaluation of the association between the incidence and severity of adenomatous proliferations and a microbiological signature has been studied, particularly at duodenal level in operated patient.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years
* Non-opposition obtained
* Prophylactic colectomy for at least 2 years in the context of APC-related familial adenomatous polyposis with ileorectal or ileoanal anastomosis
* Included in the national POLYPOSE database
* Regular endoscopic follow-up with upper and lower GI endoscopy at Hôpital Edouard Herriot or Hôpital de la Croix-Rousse
* Having performed at least 2 endoscopies as part of follow-up

Exclusion Criteria:

* Antibiotic therapy within 2 months prior to stool sampling
* Taking probiotics for less than 1 month
* Person deprived of liberty by judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with proven familial adenomatous polyposis genetically operated (total colectomy with ileoanal or ileorectal anastomosis), included in the national POLYPOSE database and with regular endoscopic follow-up with upper and lower GI endoscopy at Hôpital Edouard Herriot, Lyon, France or Hôpital de la Croix-Rousse, Lyon, France
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-12-17 (Actual); Primary Completion 2027-03-17 (Estimated); Study Completion 2027-05-17 (Estimated)

PRIMARY OUTCOMES:
Fecal microbiota composition | Within 48 hours of endoscopy
  Analysis of fecal microbiota composition as a function of the cumulative number of reservoir (rectum or ileal) adenomas treated over 3 consecutive endoscopies

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hôpital Edouard Herriot, Lyon, France
  - Hôpital de la Croix Rousse, Lyon, France